CLINICAL TRIAL: NCT06437483
Title: Effects of Sustained Natural Apophyseal Glides Combined With Kinesiotaping in Patients With Chronic Mechanical Neck Pain: A Randomised Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/7
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: In this study, participants are blinded to their assigned treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Participants in this group will receive Sustained Natural Apophyseal Glides followed by Kinesiotaping in addition to the conventional treatment. This arm of the study will assess the synergistic effects of SNAGs and kinesiotape.
  Interventions: Procedure: Sustained Natural Apophyseal Glides; Procedure: Kinesiotaping; Procedure: Conventional Treatment
- Group B (Active Comparator): Participants in group B will receive Sustained Natural Apophyseal Glides along with the conventional treatment.
  Interventions: Procedure: Sustained Natural Apophyseal Glides; Procedure: Conventional Treatment

INTERVENTIONS:
Procedure: Sustained Natural Apophyseal Glides — SNAGs:
  Therapist will apply an antero-superior accessory glide to the superior spinous process of the involved motion segment (between C3 to C7) by pushing it towards the direction of eyeball at approximately a 45 degree angle, using the thumb. The other thumb will reinforce the glide. Painless accessory glide will be maintained and subject will slowly turn their head towards the painful or restricted side (that elicited symptoms) and sustain the position for a few seconds. In case of symptom-free, the subject will apply overpressure at the end of restricted range of motion. The glide will be maintained till the head returns to the midline.
  Each session will consist of three sets of six to ten repetitions.
Procedure: Kinesiotaping — Kinesiotaping (KT):
  Subject will be in comfortable sitting position. Neck of the subject will be thoroughly cleaned with alcohol and sterile gauze pads before the application of Kinesiotape.The layers of KT will be applied in the form of two strips i.e. "Y strip" and "I strip". and applied over the neck in a position of cervical flexion and contralateral rotation and, pasted up and over either ridge of the spine covering the cervical muscles.It extends from T1-T2 to either side of C1-C2.The second layer is I-strip:The overlaying I-strip will be placed perpendicular to the Y-strip, It will be stretched from the both ends, and the middle portion of the tape will be applied first after which tension is released and ends are applied without tension.
  Arms: Group A
Procedure: Conventional Treatment — Hot pack (moist heat) and TENS will be applied, each for 10 minutes.

SUMMARY:
This study is a randomized controlled trial and its purpose is to determine the combined effects of sustained natural apophyseal glides and kinesiotaping on pain, range of motion and neck disability in patients with chronic mechanical neck pain.

DETAILED DESCRIPTION:
This study aims to determine the combined effects of sustained natural apophyseal glides and kinesiotaping in chronic mechanical neck pain patients of age range 18-40. Outcome variables are pain, range of motion and functional disability of neck which will be determined by using the following respective data collection tools:

1. Numeric pain rating scale
2. Inclinometer
3. Neck Disability Index

Participants of interest will be approached and explained about the research. They will be randomly allocated in to two groups. Informed written consent will be taken. The intervention protocol will be comprised of six sessions over a 2-week period (3 sessions per week on alternate days). Outcome measures will be assessed at baseline and after 2 weeks. Data will be analyzed and interpreted using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical Neck Pain
* Age range: 18-40 years
* Both males and females
* Having pain from at least last 3 months (chronic)
* Pain score greater than 3 on NPRS
* Pain and limitation on neck moverment

Exclusion criteria :

* Recent surgery of spine, Temporomandibular joint or shoulder in the previous 12 months.
* Open wound around neck.
* History of traumatic injuries or fractures in the cervical spine.
* History of neurological and cardiac pathologies.
* History of some serious pathologies (e.g., malignancy, inflammatory disorder etc.).
* History of cervical or shoulder neurological movement disorder.
* Cervical spondylolisthesis, cervical radiculopathy, and spinal stenosis.
* Vascular syndromes such as basilar insufficiency.
* Diagnosed psychiatric disorders such as anxiety and depression.
* Interventions including medications, exercise or physical therapy in the last 3 months.
* Any other condition that contraindicates kinesiotaping such as skin sensitivity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  It will be documented by using Numeric Pain Rating Scale (NPRS) which is a self- rated scale of 0-10 points where the participants rate their pain verbally or in writing."0" shows no pain whereas "10" represents worst pain. According to guidelines, NPRS scale categorizes pain into no pain (0), mild pain (1-3), moderate pain (4-7) and severe pain (8-10).
Cervical Range of Motion | 2 weeks
  The range of motion for flexion, extension, and side bending will be documented using a Inclinometer, positioned on the vertex of the head. For rotation, it will be placed on the forehead. Inclinometer demonstrates good Intraclass Correlation Coeffecient (ICC) value of 0.770-0.982.
Functional Disability of Neck | 2 weeks
  It will be documented by using Neck Disability Index (NDI) which consists of 10 questions addressing various aspects of neck functions to assess the impact of neck pain on a person's daily life. A total score ranges between 0 and 50 with higher scores indicating a high level of disability. Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability). All sections are then totaled.The scores on NDI are typically classified as: 0-4 (no disability), 5-14 (mild disability), 15-24 (moderate disability), 25-34 (severe disability), above 34 (complete disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan